CLINICAL TRIAL: NCT00669942
Title: A Randomized, Double Blind, Placebo-controlled, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of AIN457 in Rheumatoid Arthritis Patients With Pharmacodynamics Assessed in an Expanded Cohort at the Maximum Tolerated Dose
Brief Title: Double Blind, Placebo-controlled, Study of the Safety, Tolerability and Pharmacokinetics of AIN457 in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CAIN457A2101
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (12):
- Part 1 - AIN457A 0.3 mg/kg (Experimental): AIN457A 0.3 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - AIN457A 1.0 mg/kg (Experimental): AIN457A 1.0 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - AIN457A 3.0 mg/kg (Experimental): AIN457A 3.0 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - AIN457A 10 mg/kg (Experimental): AIN457A 10.0 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - Placebo (Placebo Comparator): Placebo to AIN457A was administered intravenously as a single dose.
  Interventions: Drug: Placebo
- Parts 2 and 3 - AIN457A 1.0 mg/kg (Experimental): AIN457A 1.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Biological: AIN457
- Parts 2 and 3 - AIN457A 3.0 mg/kg (Experimental): AIN457A 3.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Biological: AIN457
- Parts 2 and 3 - AIN457A 10 mg/kg (Experimental): AIN457A 10.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Biological: AIN457
- Parts 2 and 3 - Placebo (Placebo Comparator): Placebo to AIN457A was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Drug: Placebo
- Part 1 - Healthy Volunteers - AIN457A 3 mg/kg (Experimental): AIN457A 3.0 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - Healthy Volunteers - AIN457A 10 mg/kg (Experimental): AIN457A 10 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - Healthy Volunteers - Placebo (Placebo Comparator): Placebo to AIN457A was administered intravenously as a single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AIN457 — AIN457A is a fully human recombinant IgG1 antibody that targets and neutralizes IL-17A.
  Arms: Part 1 - AIN457A 0.3 mg/kg; Part 1 - AIN457A 1.0 mg/kg; Part 1 - AIN457A 10 mg/kg; Part 1 - AIN457A 3.0 mg/kg; Part 1 - Healthy Volunteers - AIN457A 10 mg/kg; Part 1 - Healthy Volunteers - AIN457A 3 mg/kg; Parts 2 and 3 - AIN457A 1.0 mg/kg; Parts 2 and 3 - AIN457A 10 mg/kg; Parts 2 and 3 - AIN457A 3.0 mg/kg
Drug: Placebo — Placebo to AIN457
  Arms: Part 1 - Healthy Volunteers - Placebo; Part 1 - Placebo; Parts 2 and 3 - Placebo

SUMMARY:
Evaluate the safety, tolerability and pharmacokinetics of AIN457 when administered as a single dose (intravenous infusion) in patients with active rheumatoid arthritis in combination with a stable dose of methotrexate. And to compare efficacy on the dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with active rheumatoid arthritis in combination with a stable dose of methotrexate aged 18-75 years may participate in this trial.
* Post menopausal or surgically sterile female patients are allowed. Women of child-bearing potential may participate if they are on a stable dose of methotrexate and if they are practicing effective contraception for at least 6 months prior to screening, willing to use 2 forms of contraception, including at least 1 barrier method during the study and for at least 2 months following the completion/discontinuation of the study.
* Patients must have a diagnosis of active rheumatoid arthritis of stages I, II or III (ACR 1987 revised classification for criteria for RA). Disease duration of at least 6 months prior to randomization is essential;

Exclusion Criteria:

* Current treatment with anti-TNF-α or anti IL-1 therapy (or other biological therapy).
* Patients with congestive heart failure or poorly controlled diabetes mellitus (HbA1c value ≥10%).
* Presence of any major chronic inflammatory autoimmune diseases like psoriasis, psoriatic arthritis, spondyloarthropathy, inflammatory bowel disease or SLE that can mimic rheumatoid arthritis diagnosis or that can interfere with efficacy evaluation in the study.
* History of renal trauma, glomerulonephritis or patient with one kidney.
* Pregnant or breastfeeding women will be excluded.
* A positive tuberculin skin test.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Principal Investigator — Novartis investigator site
Locations (23):
- United States (12):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Bend, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Merksem
- Germany (3):
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, München
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Guadalajara

REFERENCES:
- [Derived] Hueber W, Patel DD, Dryja T, Wright AM, Koroleva I, Bruin G, Antoni C, Draelos Z, Gold MH; Psoriasis Study Group; Durez P, Tak PP, Gomez-Reino JJ; Rheumatoid Arthritis Study Group; Foster CS, Kim RY, Samson CM, Falk NS, Chu DS, Callanan D, Nguyen QD; Uveitis Study Group; Rose K, Haider A, Di Padova F. Effects of AIN457, a fully human antibody to interleukin-17A, on psoriasis, rheumatoid arthritis, and uveitis. Sci Transl Med. 2010 Oct 6;2(52):52ra72. doi: 10.1126/scitranslmed.3001107. PMID 20926833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1: single dose escalation - sequential cohorts of patients and healthy volunteers received AIN457A or placebo. Part 2: multiple dose escalation - sequential cohorts of patients received 2 doses of AIN457A or placebo. Part 3: patients received 2 doses of AIN457 10 mg/kg (or the maximum tolerated dose) or placebo.
Pre-assignment Details: In parts 1 and 2, participants were randomized 3:1 to receive AIN457A or placebo. In part 3, participants were randomized 1:1 to receive AIN457A or placebo.
Period: Part 1
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg | Part 1 - Healthy Volunteers - Placebo
Started | 6 | 6 | 6 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Parts 2 and 3
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg | Part 1 - Healthy Volunteers - Placebo
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 26 | 26 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 24 | 23 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Healthy Volunteers
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg | Part 1 - Healthy Volunteers - Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg | Part 1 - Healthy Volunteers - Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 26 | 26 | 3 | 3 | 2 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (8.04) | 58.8 (13.61) | 51.2 (9.50) | 63.2 (9.45) | 57.8 (3.41) | 60.8 (8.66) | 56.0 (12.00) | 49.9 (8.53) | 49.8 (15.19) | 26.7 (10.02) | 22.3 (2.31) | 42.5 (10.61) | 46.07 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 5 | 7 | 5 | 3 | 19 | 20 | 0 | 0 | 1 | 75
  Male | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 7 | 6 | 3 | 3 | 1 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Parts 2 and 3 Participants Who Achieved American College of Rheumatology Response of 20 (ACR20)
Description: Clinical response to treatment was assessed according to ACR20 criteria. A participant was defined as an ACR20 responder if the following 3 conditions were met: 1) ≥20% improvement in the number of tender joints, 2) ≥20% improvement in the number of swollen joint and 3) ≥20% improvement in three of the following five domains: patient global assessment, physician global assessment, patient pain assessment, health assessment questionnaire (HAQ) and acute phase reactant.
Time Frame: Day 43
Population: The analysis was performed on the 10 mg and placebo treatment arms of the parts 2 and 3 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo
Number analyzed (Participants) | 26 | 26
percentage of participants | 46 | 27

2. Primary Outcome: Pharmacokinetics (PK) of AIN457: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part 1 Participants
Description: Serum samples were collected pre-dose and 0.5, 2, 4, 7, 12 and 24 hours post infusion on day 1, and on days 2, 5, 8, 15, 22, 29, 36, 43, 57, 71, 85, 99 and 113.
Time Frame: Day 113
Population: Part 1 participants who received AIN457A at 0.3 mg/kg, 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis. One participant in the 0.3 mg/kg arm was not analyzed due to an atypical PK profile.
Measure: Median (Full Range); unit: day
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6
day | 0.09028 [0.0833 to 0.167] | 0.08472 [0.0813 to 0.167] | 0.1253 [0.0806 to 0.167] | 0.1260 [0.0833 to 0.990]

3. Primary Outcome: PK of AIN457: Observed Maximum Serum Concentration Following Drug Administration (Cmax) in Part 1 Participants
Description: Serum samples were collected pre-dose and 0.5, 2, 4, 7, 12 and 24 hours post infusion on day 1, and on days 2, 5, 8, 15, 22, 23, 26, 29, 36, 43, 57, 71, 85, 99 and 113. On day 22, samples were collected pre-dose and 0.5, 1, 2, 4, 7 and 24 hours post infusion.
Time Frame: Day 113
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6
ug/mL | 8.772 (1.8020) | 35.22 (18.755) | 70.95 (9.9472) | 211.8 (36.837)

4. Primary Outcome: PK of AIN457: Area Under the Serum Concentration-time Cure From Time Zero to the Time of Last Quantifiable Concentration (AUClast), Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf) in Part 1 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6
day*ug/mL
  AUCinf | 141.3 (48.781) | 430.7 (48.281) | 1148 (330.89) | 4080 (768.87)
  AUClast | 132.7 (42.824) | 415.6 (42.793) | 1097 (291.59) | 3936 (697.65)

5. Primary Outcome: PK of AIN457: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz) in Part 1 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Liters | 7.043 (2.0197) | 6.756 (2.2186) | 6.506 (0.83822) | 6.699 (0.83967)

6. Primary Outcome: PK of AIN457: Systemic Clearance From Serum Following Intravenous Administration (CL) in Part 1 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Liters/day | 0.2249 (0.11196) | 0.2110 (0.064415) | 0.2077 (0.080880) | 0.1999 (0.049375)

7. Primary Outcome: PK of AIN457: Terminal Elimination Half-life (T1/2) in Part 1 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Part 1 participants who received AIN457A at 0.3 mg/kg, 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
day | 23.21 (6.8285) | 22.27 (2.8478) | 23.47 (5.7952) | 23.94 (4.2566)

8. Primary Outcome: Pharmacokinetics PK of AIN457: Tmax in Parts 2 and 3 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Parts 2 and 3 participants who received AIN457A at 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Median (Full Range); unit: day
Arm/Group | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 26
day | 21.08 [0.167 to 21.2] | 21.08 [20.1 to 21.3] | 21.09 [0.0736 to 21.4]

9. Primary Outcome: Pharmacokinetics PK of AIN457: Cmax in Parts 2 and 3 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Parts 2 and 3 participants who received AIN457A at 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 26
ug/mL | 23.54 (3.1588) | 97.78 (15.543) | 322.2 (96.719)

10. Primary Outcome: Pharmacokinetics PK of AIN457: AUClast and AUCinf in Parts 2 and 3 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Parts 2 and 3 participants who received AIN457A at 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 26
day*ug/mL
  AUCinf | 808.6 (251.01) | 2843 (481.49) | 8371 (2505.8)
  AUClast | 746.4 (209.20) | 2704 (467.60) | 7815 (2102.0)

11. Primary Outcome: Pharmacokinetics PK of AIN457: Vz in Parts 2 and 3 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Parts 2 and 3 participants who received AIN457A at 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 26
Liter | 6.514 (1.1542) | 6.062 (1.0189) | 6.382 (1.1336)

12. Primary Outcome: Pharmacokinetics PK of AIN457: CL in Parts 2 and 3 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Parts 2 and 3 participants who received AIN457A at 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 26
Liters/day | 0.1834 (0.042822) | 0.1775 (0.034075) | 0.1994 (0.063454)

13. Primary Outcome: Pharmacokinetics PK of AIN457: T1/2 in Parts 2 and 3 Participants
Description: as for outcome 3
Time Frame: Day 113
Population: Parts 2 and 3 participants who received AIN457A at 1 mg/kg, 3 mg/kg or 10 mg/kg were included in this analysis.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Parts 2 and 3 - AIN457A 1.0 mg/kg | Parts 2 and 3 - AIN457A 3.0 mg/kg | Parts 2 and 3 - AIN457A 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 26
Day | 25.60 (6.3100) | 23.89 (3.2335) | 23.68 (6.3048)

14. Secondary Outcome: Percentage of Parts 2 and 3 Participants Who Achieved ACR50 and ACR70
Description: Clinical response to treatment was assessed according to ACR50 and ACR70 criteria. A participant was defined as an ACR50 or ACR70 responder if the following 3 conditions were met: 1) improvement of ≥50% or ≥ 70%, respectively, in the number of tender joints, 2) improvement of ≥50% or ≥ 70%, respectively, in the number of swollen joints and 3) improvement of ≥50% or ≥ 70%, respectively, in three of the following five domains: patient global assessment, physician global assessment, patient pain assessment, health assessment questionnaire (HAQ) and acute phase reactant
Time Frame: Day 43
Population: The analysis was performed on the 10 mg and placebo treatment arms of the parts 2 and 3 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo
Number analyzed (Participants) | 26 | 26
Percentage of participants
  ACR50 | 27 | 15
  ACR70 | 8 | 8

15. Secondary Outcome: Disease Activity Score (DAS28) of Parts 2 and 3 Participants
Description: The DAS28 is a composite score based on tender and swollen joint counts, C reactive protein (CRP) concentrations, and the participant's global disease activity based on a visual analogue scale (VAS). The tender joint count (based on 28 joints) was calculated by scoring several different aspects of tenderness as assessed by pressure and joint manipulation on physical examination. The information on various types of tenderness was then collapsed into a single tender versus non-tender dichotomy, and the number of joints that were classified as tender was recorded. The swollen joint count was calculated in the same manner. For CRP concentrations, blood samples were collected and sent to a central laboratory for assessment. For the VAS assessment, the participant used a 100 mm horizontal VAS to assess the severity of his or her arthritis where 0 = none and 100 = most severe. DAS28 scores range from <2.6 (disease remission) to >5.1 (high disease activity).
Time Frame: Day 43
Population: The analysis was performed on the 10 mg and placebo treatment arms of the parts 2 and 3 participants.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Parts 2 and 3 - AIN457A 10 mg/kg | Parts 2 and 3 - Placebo
Number analyzed (Participants) | 25 | 23
scores on a scale | 4.306 (1.4787) | 4.598 (1.2618)

ADVERSE EVENTS:
Groups:
- Parts 2 and 3 - AIN457 1.0 mg/kg: AIN457A 1.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
- Parts 2 and 3 - AIN457 3.0 mg/kg: AIN457A 3.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
- Parts 2 and 3 - AIN457 10 mg/kg: AIN457A 10.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
Arm/Group | Part 1 - AIN457A 0.3 mg/kg | Part 1 - AIN457A 1.0 mg/kg | Part 1 - AIN457A 3.0 mg/kg | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 2 and 3 - AIN457 1.0 mg/kg | Parts 2 and 3 - AIN457 3.0 mg/kg | Parts 2 and 3 - AIN457 10 mg/kg | Parts 2 and 3 - Placebo | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg | Part 1 - Healthy Volunteers - Placebo | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/6 | 0/6 | 0/8 | 0/6 | 1/6 | 0/26 | 2/26 | 0/3 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 5/6 | 2/6 | 4/8 | 5/6 | 4/6 | 19/26 | 13/26 | 1/3 | 1/2 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - AIN457A 0.3 mg/kg (N=6) | Part 1 - AIN457A 1.0 mg/kg (N=6) | Part 1 - AIN457A 3.0 mg/kg (N=6) | Part 1 - AIN457A 10 mg/kg (N=6) | Part 1 - Placebo (N=8) | Parts 2 and 3 - AIN457 1.0 mg/kg (N=6) | Parts 2 and 3 - AIN457 3.0 mg/kg (N=6) | Parts 2 and 3 - AIN457 10 mg/kg (N=26) | Parts 2 and 3 - Placebo (N=26) | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg (N=3) | Part 1 - Healthy Volunteers - Placebo (N=2) | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg (N=3)
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - AIN457A 0.3 mg/kg (N=6) | Part 1 - AIN457A 1.0 mg/kg (N=6) | Part 1 - AIN457A 3.0 mg/kg (N=6) | Part 1 - AIN457A 10 mg/kg (N=6) | Part 1 - Placebo (N=8) | Parts 2 and 3 - AIN457 1.0 mg/kg (N=6) | Parts 2 and 3 - AIN457 3.0 mg/kg (N=6) | Parts 2 and 3 - AIN457 10 mg/kg (N=26) | Parts 2 and 3 - Placebo (N=26) | Part 1 - Healthy Volunteers - AIN457A 3 mg/kg (N=3) | Part 1 - Healthy Volunteers - Placebo (N=2) | Part 1 - Healthy Volunteers - AIN457A 10 mg/kg (N=3)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.